CLINICAL TRIAL: NCT04498325
Title: A Phase I and Pilot Study Evaluating the Effect of NT-I7, a Long Acting Interleukin-7, to Increase Lymphocyte Counts and Enhance Immune Clearance of SARS-CoV-2
Brief Title: Evaluating the Effect of NT-I7, a Long Acting Interleukin-7, to Increase Lymphocyte Counts and Enhance Immune Clearance of SARS-CoV-2 (COVID-19)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal investigator is leaving the institution.
Sponsor: Washington University School of Medicine (Other)
Collaborators: NeoImmuneTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202009065
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — efineptakin alfa; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The study will open as a phase I study to test three different dose levels of NT-I7. Once a safe tolerated dose is established, the pilot portion of the study will be activated wherein participants will be randomized on a 1:1 basis to receive a single injection of NT-I7 (at the safe tolerated dose) or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The clinicians, participants, and clinical research coordinators will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NT-I7 (Phase I) (Experimental): * In the phase I study, 3 dose levels of NT-I7 are planned. Dosing will be staggered such that there will be a minimum of 72 hours between the dosing of one participant and the dosing of the next participant
  * NT-I7 will be given by intramuscular injection on Day 0
  * Participants will also be given standard of care treatment for COVID-19
  Interventions: Drug: NT-I7; Procedure: Blood for research purposes; Procedure: Blood for pharmacokinetic samples; Procedure: Nasopharyngeal, oropharyngeal, or saliva swab; Procedure: Blood for anti-drug antibody (ADA)
- NT-I7 (Pilot) (Experimental): * NT-I7 (dose determined by Phase I portion of study) will be given by intramuscular injection on Day 0
  * Participants will also be given standard of care treatment for COVID-19
  Interventions: Drug: NT-I7; Procedure: Blood for research purposes; Procedure: Nasopharyngeal, oropharyngeal, or saliva swab; Procedure: Blood for anti-drug antibody (ADA)
- Placebo (Pilot) (Placebo Comparator): * Placebo will be given by intramuscular injection on Day 0
  * Participants will also be given standard of care treatment for COVID-19
  Interventions: Drug: Placebo; Procedure: Blood for research purposes; Procedure: Nasopharyngeal, oropharyngeal, or saliva swab; Procedure: Blood for anti-drug antibody (ADA)

INTERVENTIONS:
Drug: NT-I7 — Supplied by study
  Arms: NT-I7 (Phase I); NT-I7 (Pilot)
Drug: Placebo — Supplied by study
  Arms: Placebo (Pilot)
Procedure: Blood for research purposes — Prior to injection (Day 0), Day 7, and Day 14
Procedure: Blood for pharmacokinetic samples — -Phase I only: 1-2 hours prior to dosing, 6 hours after dosing, 24 hours after dosing, Day 7, Day 14, and Day 21
  Arms: NT-I7 (Phase I)
Procedure: Nasopharyngeal, oropharyngeal, or saliva swab — -Prior to study treatment, Day 4(optional), Day 7, and Day 14
Procedure: Blood for anti-drug antibody (ADA) — Baseline, Day 7, Day 14, Day 21, Day 60, and Day 90. Participants with ADA positivity on Day 90 will be monitored every 90 days until antibody level returns to baseline

SUMMARY:
Lymphopenia is common in patients with COVID-19 and is associated with worse clinical outcomes. NT-I7 is a long-acting human interleukin-7 (IL-7) that has been shown to increase absolute lymphocyte count (ALC) and CD4+ and CD8+ T cell counts with a well-tolerated safety profile in humans. In this study, patients who have tested positive for SARS-CoV-2 by PCR testing without severe disease and with ALC <1500 cells/mm3 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Tested PCR positive for SARS-CoV-2by nasopharyngeal swab, oropharyngeal swab, or saliva.
* Mild COVID-19, defined as WHO Ordinal Scale <4 .
* Respiratory rate < 20 bpm, HR < 90 bpm, and SpO2 > 93% on room air at sea level.
* Absolute lymphocyte count (ALC) < 1500 cells/mm3 at the time of screening.
* AST/ALT ≤ 3.0 x ULN, total bilirubin ≤ 1.5 x ULN (except if due to Gilbert's syndrome).

  -≥ 18 years of age.
* First day of treatment must be no more than 10 days from onset of COVID-19 symptoms.
* Must be willing to be closely monitored in the hospital or in an alternate setting (e.g. clinical trial unit) for at least the first 7 days (±2 days allowed) following NT-I7/placebo injection.
* Individuals of reproductive potential must agree to either abstinence or use of at least one study-approved form of contraception when engaging in sexual activities that can result in pregnancy from the time of screening through 60 days for female and 120 days for male after study agent administration. Acceptable forms of contraception for this study are male or female condoms, diaphragms or cervical caps with a spermicide, or non-hormonal intrauterine devices.
* Patients with factors or concomitant illness associated with higher risk of mortality due to COVID-19 (such as older age, hypertension, diabetes, and/or COPD) are eligible.
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Receiving any other investigational agents which may affect patient's lymphocyte counts. Note: There is no evidence that chloroquine or hydroxychloroquine could affect lymphocyte counts. Thus, chloroquine or hydroxychloroquine use is not an exclusion criteria for this study. Additionally, it is permissible for potential participants to have received investigational or off-label agents for COVID-19 prior to or during study participation.
* Pregnant or breastfeeding women are excluded from this study because NT-I7 has not been evaluated regarding its potential for teratogenic or abortifacients effects. There is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drug; therefore, breastfeeding should be discontinued if the mother is treated with NT-I7.
* Transferred from ICU to the floor.
* Requiring dialysis.
* Shortness of breath or known hypoxia (defined as PaO2/FiO2 ≤ 300 mmHg), or signs of serious lower airway disease.
* Evidence of ARDS, SIRS/shock, or cardiac failure.
* Elevated inflammatory markers such as CRP > 2 x ULN, LDH > 2 x ULN, D-dimer > 2 x ULN, ferritin > ULN, or IL-6 > ULN (when available).
* Any established diagnosis of autoimmune disease requiring systemic treatment EXCEPT for vitiligo or endocrine disease (such as diabetes, thyroid disease, and adrenal disease) controlled by replacement therapy.
* Receipt of live attenuated vaccine within 30 days before the study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), Zoster, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Safe and tolerable dose of NT-I7 (Phase I only) | Completion of DLT assessment window of Phase I portion of study (estimated to be 8 months)
  * The safe tolerated dose is defined as the dose level immediately below the dose level at which 1 patient of a cohort of 3 patients experiences dose-limiting toxicity within 14 days after administration of NT-I7
  * Dose limiting toxicities (DLT) are defined as:
    * A serious adverse event that is at least possibly related to NT-I7
    * A grade 3 or higher adverse event that is at least possibly related to NT-I7 (excluding injection site swelling, irritation or discomfort)
    * A clinically significant lab abnormality that is at least possibly related to NT-I7
Percent change in absolute lymphocyte count (ALC) | From baseline to Day 14

SECONDARY OUTCOMES:
Percent change in absolute lymphocyte count (ALC) | From baseline through Day 21
Change in SARS-CoV-2 viral load | From baseline to Day 7
  -Using PCR from nasopharyngeal swab, oropharyngeal swab or saliva
Change in SARS-CoV-2 viral load | From baseline to Day 14
  -Using PCR from nasopharyngeal swab, oropharyngeal swab or saliva
COVID-19 Symptom severity as measured by WHO Ordinal Scale for clinical improvement | From baseline, day 7, day 14, and day 21
Time to resolution of COVID-19 symptoms | From baseline through Day 21
Incidence of treatment-emergent adverse events | From baseline through Day 21
  -A treatment emergent adverse event (TEAE) is defined as any event that begins or worsens on or after date of first dose of study treatment.
Number of participants by PCR result status (positive or negative) | -From baseline to Day 7
  -If quantitative PCR is not available
Number of participants by PCR result status (positive or negative) | From baseline to Day 14
  -If quantitative PCR is not available

CONTACTS AND LOCATIONS:
Overall Officials: Jian Campian, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu